CLINICAL TRIAL: NCT01062204
Title: A Randomized Comparison Study of a Flexible HydrogelNanoparticle Wound Dressing (Altrazeal) Versus a Sodium Carboxymethylcellulose Dressing (Aquacel Ag) as Dressings for Partial Thickness Skin Graft Donor Sites
Brief Title: Altrazeal™ Versus Aquacel® Ag for Partial Thickness Skin Donor Sites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ULURU Inc. (Industry)
Responsible Party: Brett Arnoldo, MD, UTSW Medical Center, Department of Surgery
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-6U1102
Record Dates: First submitted 2010-02-02; First posted 2010-02-04 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Partial-thickness Skin Donor Sites
Keywords: Skin Graft donor sites

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Altrazeal — Sterile, odorless, crystalline white powder consisting of flakes of freeze dried HEMA and HPMA polymers. For application, the powder is distributed to the surface of the wound or burn where it forms a moist, flexible film and adheres to the surface of the wound.
Device: Aquacel Ag — Textile fiber made from sodium carboxy-methylcellulose containing 1.2% silver in ionic form.

SUMMARY:
The primary objective of the study is to evaluate the time to wound healing in skin graft donor sites with a new treatment (Altrazeal dressing) compared to standard of care treatment (Aquacel Ag- Carboxymethylcellulose dressing) in partial thickness skin graft donor sites.

DETAILED DESCRIPTION:
This is a single center, randomized, therapeutic exploratory study to monitor wound healing with the new AltrazealTM flexible hydrogel nanoparticle dressing compared to the existing treatment standard (Aquacel ® AG sodium carboxymethylcellulose dressing) in patients with at least two skin graft donor sites. 40 patients with at least 2 skin graft donor sites, ranging in age from 3 and 85 years, will be enrolled. Children (age 3 to 16 inclusive) will be included in the patient population if possible, but should not exceed 50% of all patient enrolled. Researchers will first identify the skin donor sites (A and B) for each patient and take baseline digital images and measurements immediately following surgery (Day 1). Trained personnel will apply the dressings provided by the Sponsor for and labeled as A or B by the Sponsor in a random fashion. Typical meticulous wound care and adequate analgesic medical coverage will be provided for the duration of the study. Both the patient and medical staff will be trained on instructions for use of each dressing. The patients will be monitored daily as part of standard procedure while they are in the in-patient setting. If and when patients move to the out-patient setting, they will continue to be monitored at least every-other-day at the study center. On each day (in-patient) or every-other-day (outpatient), the physician will determine whether each skin graft donor site has healed per standard care guidelines (i.e. > 95% re-epithelization), and pain and adverse events will be monitored. The last study visit will be on Day 24 or on the day when both wounds have been assessed as "healed", whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient is between the ages of 3 and 85 Note: In order to maintain a broad representation of ages, no more than 50% of the patients enrolled in the study should be between the ages of 3 and 16, inclusive.
2. Patient is in general good health
3. Patient has two independent skin donor sites of approximately the same dimensions.
4. Patient is willing and able to cooperate with the protocol for duration of study.
5. Patient is capable of providing informed consent and HIPAA authorization
6. Ability to read and speak either English or Spanish

Exclusion Criteria:

1. Male or female patient is less than 3 years of age or more than 85 years of age
2. Patient has acutely infected wounds
3. Patient has wounds with surrounding cellulites
4. Patient has a history of hypersensitivity to any components of either the nanoparticle or sodium carboxymethylcellulose dressing, or any known sensitivities to other hydrogel bandage treatments
5. Patient has a concurrent clinical condition, which in the judgment of the Investigator could either pose a health risk to the patient while participating in this study, or could potentially influence the outcome of the study;
6. Patient has history of poor wound healing or any skin/immune system condition that would increase likelihood of wound irritation, infection or increase chance of early termination
7. Patient is unable to communicate or to cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function.

Ages: 3 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Time to wound healing (re-epithelialization), in days assessed by the physician according to the study center's Standard of Care, for each wound dressing. | 24 days

SECONDARY OUTCOMES:
Patient's comfort | 24 days
Patient's pain | 24 days
Infections | 24 days

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States